CLINICAL TRIAL: NCT04075058
Title: A Phase III Randomized Study Comparing Two Adjuvant Hypofractionated Radiation Schedules in Patients With Breast Cancer
Brief Title: Hypofractionated Radiation Therapy in Patients With Breast Cancer
Acronym: HRBC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Budhi Singh Yadav, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRBC
Record Dates: First submitted 2015-10-26; First posted 2019-08-30 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer; hypofractionated radiotherapy; Hypofractionated radiation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study (Experimental): Patients with breast cancer post mastectomy or after breast conservative surgery to be treated with a hypofractionated radiotherapy dose of 34Gy in 10 fractions over 2 weeks.
  Interventions: Radiation: Hypofractionated Radiation therapy
- Control (Active Comparator): Patients with breast cancer post mastectomy or after breast conservative surgery to be treated with a hypofractionated radiotherapy dose of 35Gy in 15 fractions over 3 weeks
  Interventions: Radiation: Hypofractionated Radiation therapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation therapy

SUMMARY:
The investigators at PGIMER have been practicing hypofractionation radiotherapy with a dose of 35Gy/15#/3wks to the chest wall in post mastectomy and 40Gy/16#/3wks in breast conservation in breast cancer patients for the last 4 decades. It is also a routine practice in UK and few centers in Canada. Hypofractionation reduces treatment time to half while maintaining cosmesis and gives control rates equal to conventional fractionation. As breast cancer is a leading cancer in females and radiation therapy is an important part of its local management, hypofractionation help the radiation centers worldwide to meet the growing need for radiation in breast cancer, particularly in developing countries where resources are limited. It also reduces the financial burden on the patient and family. In this study the investigators want to reduce the treatment duration from 3 weeks to 2 weeks. The study will include 1000 patients, 500 in each arm, with breast cancer post mastectomy or after breast conservative surgery to be treated with a radiotherapy dose of 34Gy in 10 fractions over 2 weeks in the study arm and 35Gy in 15 fractions over 3 weeks in the control arm. The primary endpoint of the study will be ipsilateral local tumour control. Secondary endpoints will be early and late adverse effects in normal tissues, quality of life, contralateral primary tumours, regional and distant metastases and survival.

DETAILED DESCRIPTION:
Patients to be included in this study will be pre-operatively staged according to American Joint Committee on Cancer (AJCC) 7th edition, International Union against cancer ( which uses TNM staging ) as stage I-III of breast carcinoma. Total 500 patients of histologically proven post lumpectomy/mastectomy cases of carcinoma breast suitable for radiotherapy will be enrolled in this study. Patients would be evaluated at the Department of Radiotherapy PGIMER, Chandigarh by doing a thorough clinical examination followed by routine investigations which will include hemogram, liver function tests, kidney function tests, chest X-ray. Patients will be treated by standard rectangular tangential fields.

ELIGIBILITY:
Inclusion Criteria:

* Invasive carcinoma of the breast
* Breast conservation surgery or mastectomy
* Axillary staging &/or dissection
* Complete microscopic excision of primary tumour
* pT1-3 pN0-2 M0 disease
* Written informed consent
* Able to comply with follow up

Exclusion Criteria:

* Past history of malignancy except (i) basal cell skin cancer and CIN cervix uteri or (ii) non-breast malignancy allowed if treated with curative intent and at least 5 years disease free
* Contralateral breast cancer, including DCIS, irrespective of date of diagnosis
* Breast reconstruction using implants
* Concurrent cytotoxic chemotherapy (sequential neoadjuvant or adjuvant cytotoxic therapy allowed)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1070 (Actual)
Dates: Start 2015-06; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Local Recurrence | 5 years
  Any recurrence with in the irradiated area from completion of radiation

SECONDARY OUTCOMES:
Acute skin toxicity | After 1 month of completion of radiation
  Acute toxicity will be assessed using a RTOG grading system. Assessment will be carried out weekly during radiotherapy and for 4 weeks after treatment.
Cosmetic assessment | Baseline, 1 year, 3 years, 5 years
  done using Harvard/National Surgical Adjuvant Bowel and Breast Project(NSABP)/Radiation Therapy Oncology Group(RTOG) breast cosmesis grading scale. Grading will be done as Excellent- no or minimal difference between two breasts,Good- slight difference between two breasts,Good- slight and Fair minimal difference between two breasts, Fair- obvious difference between two breasts Poor- marked difference between two breasts. Excellent/good and fair/poor will be considered better and worse outcomes, respectively.
Quality of life | 3 year, 5 year
  EORTC QLQ -30 The QLQ-C30 is composed of both multi-item scales and single-item measures, as well as five functional scales, three symptom scales, a global health status/QoL scale, and six single items.The scores must be averaged and linearly transformed to obtain a range of scores from 0 to 100, with a higher score representing a greater response level. Thus, a high score for a functional scale represents a healthy level of functioning and a high score for the global health status represents a high QoL, but a high score for the symptom scale represents a high level of symptomatology.
Quality of life | 3 year, 5 year
  EORTC QLQ-BR 23 It contains 23 items rated on a four-point scale ranging from 1 (not at all) to 4 (very much). The items assess the side effects of therapy, arm symptoms, breast symptoms, body image, and sexual function. Additionally, there are single items assessing sexual enjoyment, anxiety caused by hair loss, and future outlook. The scores range between 0-100 points. For scales evaluating function, a higher score represents a higher level of functioning. For scales evaluating symptoms, a higher score indicates more severe symptoms.
Disease free survival | 5 years, 10 years
  Time interval free from locoregional recurrence and metastasis
Overall survival | 5 years, 10 years
  From the date of diagnosis to death
Arm edema | 3 years, 5 years, 10 years
  Will be graded by measuring arm circumference 10cm above and below the medial epicondyle of humerus. Treated side will be compared with the untreated opposite side as a reference. It will be classified as none, mild, moderate and marked if there was no difference, 0.5-2cm, 2.1-3cm and >3cm difference, respectively in the circumference of the affected and normal arm.
Late effects- pain, shoulder stiffness | 3 years, 5 years, 10 years
  A four point scale(none, a little, quite a bit, very much ) will be used to asess all late effects according to the RTOG LENT SOMA scale(Cox et al, 1995).
Late effects- Brachial plexopathy | 3 years, 5 years, 10 years
  If the patient had symptoms of pain in the arm, paresthesia, numbness, weakness, or other sensory symptoms then injury to the brachial plexus will be suspected and reported as brachial plexopathy.
Late effects- Lung, cardiac | 5 years, 10 years
  Late lung and cardiac toxicity asess all late effects according to the RTOG LENT SOMA scale (Cox et al, 1995).

CONTACTS AND LOCATIONS:
Overall Officials: Budhi S Yadav, MD, Principal Investigator — PGIMER, Chandigarh, India
Locations (1):
- Dr Budhi Singh Yadav, Chandigarh, N/A = Not Applicable, India

REFERENCES:
- [Background] Yadav BS. Accelerated partial breast irradiation. Radiother Oncol. 2009 Jan;90(1):161. doi: 10.1016/j.radonc.2007.10.005. Epub 2007 Oct 25. No abstract available. PMID 17963907
- [Background] Yadav BS, Sharma SC, Patel FD, Ghoshal S, Kapoor RK. Second primary in the contralateral breast after treatment of breast cancer. Radiother Oncol. 2008 Feb;86(2):171-6. doi: 10.1016/j.radonc.2007.10.002. Epub 2007 Oct 24. PMID 17961777
- [Result] Yadav BS, Sharma SC, George P, Bansal A. Post-mastectomy radiation beyond chest wall in patients with N1 breast cancer: is there a benefit? J Cancer Res Ther. 2014 Apr-Jun;10(2):279-83. doi: 10.4103/0973-1482.136560. PMID 25022378
- [Result] Yadav BS, Sharma SC, Patel FD, Ghoshal S, Kapoor R, Kumar R. Nonbreast second malignancies after treatment of primary breast cancer. Int J Radiat Oncol Biol Phys. 2009 Apr 1;73(5):1489-92. doi: 10.1016/j.ijrobp.2008.07.004. Epub 2008 Sep 19. PMID 18804919
- [Derived] Yadav BS, Dahiya D, Gupta M, Gupta A, Oinam AS, Khare S, Irrinki S, Robert N, Sakaray YR, Nagaraj SS, Kumari R. Preliminary results of hypofractionated radiotherapy in breast cancer in Chandigarh, India: single-centre, non-inferiority, open-label, randomised, phase 3 trial. Lancet Reg Health Southeast Asia. 2024 Mar 21;24:100392. doi: 10.1016/j.lansea.2024.100392. eCollection 2024 May. PMID 38550605